CLINICAL TRIAL: NCT05054426
Title: Intravenous Methotrexate 1g/m2 as Central Nervous System Prophylaxis for High Risk Diffuse Large B Cell Lymphoma: a Prospective, Phase III, Randomized, Controlled Study
Brief Title: Intermediate Dose of IV MTX as CNS Prophylaxis for High Risk DLBCL
Acronym: NHL-011
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, YanZhang, associate professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-NHL-011
Record Dates: First submitted 2021-09-01; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Diffuse Large B Cell Lymphoma; Central Nervous System Lymphoma
Keywords: central nervous system prophylaxis; methotrexate
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intravenous MTX (Experimental): intravenous methotrexate at a dose of 1g/m2 for 4 courses
  Interventions: Drug: Methotrexate
- intrathecal MTX (Experimental): intrathecal methotrexate 10mg at a time for 4 courses
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — intravenous versus intrathecal methotrexate

SUMMARY:
Central nervous system (CNS) relapse is a devastating event of diffuse large B cell lymphoma (DLBCL). It occurs in 4%-7% of DLBCL in general and the rate is considerably higher in high-risk patients, resulting in a poor outcome.Effective methods of CNS prophylaxis have not yet been developed. Evidence for intrathecal or intravenous MTX are both controversial. In one previous study of PUMCH, IV MTX at a dose of 1g/m2 could significantly decrease the 2 year CNS relapse rate of high risk DLBCL(1.1% vs 12.1% for historic cohort, P=0.003). In current study, the investigators are aiming to confirm its efficacy through phase III study with intrathecal MTX as the controlled arm.

DETAILED DESCRIPTION:
In this prospective, phase III, multicenter, randomized, controlled study, the investigatirs aim to compare the efficacy of intravenous MTX(IV arm) at a dose of 1g/m2 with intrathecal MTX(IT arm) in terms of preventing CNS relapse. All the patients will recieve RCHOP regimen as front-line treatment of DLBCL. Patients in IV arm will recieve 4 course of IV MTX, which is incorporated into the RCHOP, naming R-MTX-CHOP regimen. Patients in IT arm will be given intrathecal MTX for 4 courses (one time for each course). 2 year CNS relapse rate is the primary endpoint while 2 year PFS, 2 year OS and safety are the secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* with high CNS risk, which was defined as involvement of more than one extranodal site, or involvement of particular extranodal sites such as bone marrow, breasts, testes, paranasal sinuses, epidural space, adrenal glands, kidney and female genital system;
* first-line treatment planned to be RCHOP
* absence of CNS involvement at presentation

Exclusion Criteria:

* primary CNS lymphoma
* already have CNS involvement at diagnosis
* primary mediastinal lymphoma, intravascular large B-cell lymphoma, DLBCL leg-type, Burkitt lymphoma, high-grade lymphomas, double expressor lymphoma
* with active infection or other malignancy
* severe liver or kidney insufficiency
* allergy to any medication we plan to use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2021-10-08 (Estimated); Primary Completion 2025-10-08 (Estimated); Study Completion 2025-10-08 (Estimated)

PRIMARY OUTCOMES:
2 year CNS relapse rate | 2 year
  CNS relapse was defined as positive CSF conventionalcytology, CSF flow cytometry, or biopsy. For those who had clinical symptoms indicating a CNS involvement and typical lesions on MRI, the investigators also considered a recurrence

SECONDARY OUTCOMES:
progression free survival | 2 year
  from diagnosis to any event including progression, relapse and death
overall survival | 2 year
  from diagnosis to death

CONTACTS AND LOCATIONS:
Overall Officials: Daobin Zhou, MD., Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking union medical college hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang W, Zhang Y, Zhang L, Yang C, Feng J, Cai H, Chen M, Cao X, Zhuang J, Zhu T, Duan M, Zhang W, Li J, Zhou D. Intravenous methotrexate at a dose of 1 g/m2 incorporated into RCHOP prevented CNS relapse in high-risk DLBCL patients: A prospective, historic controlled study. Am J Hematol. 2020 Apr;95(4):E80-E83. doi: 10.1002/ajh.25723. Epub 2020 Jan 22. No abstract available. PMID 31925808